CLINICAL TRIAL: NCT01465347
Title: Open-label Phase 1/2 (Safety Lead-in) Study of Trans Sodium Crocetinate (TSC) With Concomitant Treatment of Fractionated Radiation Therapy and Temozolomide in Newly Diagnosed Glioblastoma (GBM) Patients to Evaluate Safety and Efficacy
Brief Title: Safety and Efficacy of Trans Sodium Crocetinate (TSC) With Radiation and Temozolomide in Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP100-202
Record Dates: First submitted 2011-11-02; First posted 2011-11-04 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Glioblastoma; GBM; Glioma
Keywords: Primary brain tumor; Glioblastoma; Glioma; GBM; Radiation therapy
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — trans-sodium crocetinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TSC 0.25 mg/kg for 9 or 18 doses (Experimental): This was an open-label, sequential-cohort, dose-escalation study in two phases. Phase 1 was a safety run-in evaluating Trans Sodium Crocetinate (TSC) in 3 subjects who received 3 doses per week for 3 weeks (9 doses in total). Phase 2 engaged 56 subjects who received 3 doses per week for 6 weeks (18 doses in total). TSC was consistently dosed at 0.25mg/kg in both phases.
  Interventions: Drug: Trans Sodium Crocetinate (TSC)

INTERVENTIONS:
Drug: Trans Sodium Crocetinate (TSC) — TSC administered intravenously as a bolus injection prior to radiation therapy sessions during 6 weeks of radiotherapy.
  Other Names: TSC

SUMMARY:
This open-label study evaluated the safety and efficacy of TSC when dosed concomitantly with the standard of care (radiation therapy and temozolomide) for newly diagnosed glioblastoma in adults. All patients received TSC in the study. The objective of the study was to evaluate the effect of TSC on survival and tumor response in patients with GBM while establishing an acceptable patient risk profile.

DETAILED DESCRIPTION:
The overall objectives of this Phase 1/2 clinical study in newly diagnosed GBM patients was to evaluate the safety and tolerability, efficacy, PK profile, PFS/time to disease progression, QoL, and overall survival in adults when TSC is added to the standard of care regimen of radiation therapy and temozolomide. All patients received TSC in this study. The primary objective of the Phase 1 portion of the study was to evaluate the safety (DLT rate) and to define the dosing regimen of TSC for the larger Phase 2 study. The primary clinical endpoint was overall survival at 24 months and patients will be followed for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years of age; male or female. A patient who is 70 years of age or older may be considered for enrollment after review of patient clinical and laboratory data by the Protocol Medical Monitor.
* Histologically confirmed diagnosis of GBM.
* Contrast enhancing disease on MRI within 21 days prior to screening.
* Karnofsky score (KPS) of ≥ 60 at Screening.
* No prior RT, chemotherapy (including Gliadel wafer), immunotherapy or therapy with a biologic agent, or hormonal therapy. Glucocorticoid therapy is allowed.
* Within 2 weeks of baseline visit, hematologic and renal functions as specified: Absolute neutrophil count ≥ 1500/mm3, platelets ≥ 100,000/mm3, Hgb ≥ 9.0g/dL, creatinine ≤ 1.7mg/dl, total bilirubin ≤ 1.5mg/dL, blood urea nitrogen (BUN) within 2 times the upper limit of normal, transaminases ≤ 4 times above the upper limits of the institutional norm.
* Sexually active patients must use an acceptable method of contraception while receiving doses of study medication.
* Females of childbearing potential must have a negative serum or urine pregnancy test at screening and have additional pregnancy tests during study.

Exclusion Criteria:

* Patient who cannot undergo MRI.
* Pregnant or lactating.
* Serious concurrent infection or medical illness that would jeopardize the ability of the patient to receive study treatment with reasonable safety.
* Patient receiving concurrent chemotherapeutics or investigational agents within 30 days of baseline assessments, including gliadel wafers or gliasite application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Jones, M.D., Study Chair — Diffusion Pharmaceuticals Inc
Locations (18):
- United States (18):
  - St. Joseph's Medical Center Barrow Neurology Clinics, Phoenix, Arizona
  - University of Arkansas Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - North Shore University Hospital, Manhasset, New York
  - Forsyth Regional Cancer Center, Winston-Salem, North Carolina
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Health Science Center Memorial Hermann Medical Center, Houston, Texas
  - UVA Health Sciences Center Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Froedtert & Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Derived] Gainer JL, Sheehan JP, Larner JM, Jones DR. Trans sodium crocetinate with temozolomide and radiation therapy for glioblastoma multiforme. J Neurosurg. 2017 Feb;126(2):460-466. doi: 10.3171/2016.3.JNS152693. Epub 2016 May 13. PMID 27177177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment naive patients with a histologically confirmed diagnosis of GBM who were scheduled to receive standard-of-care radiation and temozolomide treatment per Stupp et al (2005) were enrolled in the study at 18 academic clinical sites in the U.S.
Pre-assignment Details: Open-label, historical control (Stupp et al; N Engl J Med 2005; 352: 987-996, March 10, 2005, DOI: 10.1056/NEJMoa043330); patients received standard-of-care radiation/temozolomide treatment plus Trans Sodium Crocetinate (TSC); three (3) patients completed 9 doses (phase 1) as a safety run-in followed by 56 patients who received 18 doses (phase 2).
Groups:
- TSC 0.25 mg/kg - 9 Dose Group: Phase 1: 3 weeks of TSC (9 doses in total) with concomitant RT and temozolomide for 6 weeks
- TSC 0.25 mg/kg - 18 Dose Group: Phase 2: 6 weeks of TSC (18 doses in total) with concomitant RT and temozolomide for 6 weeks
Period: Overall Study
Arm/Group | TSC 0.25 mg/kg - 9 Dose Group | TSC 0.25 mg/kg - 18 Dose Group
Started | 3 | 56
Completed | 2 | 53
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Admitted to hospice | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was the 56 patients in phase 2 given the comparison to historical control (Stupp 2005) wherein patients were treated for 6 weeks.
Arm/Group | TSC 0.25 mg/kg for 9 or 18 Doses
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 52
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 56
Count of participants [Number; unit: participants] | 56

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLTs)
Description: Number of Participants in Phase 1 with Dose Limiting Toxicities (DLTs)
Time Frame: During phase 1
Population: Dose limiting toxicities were only assessed for Phase 1 participants
Measure: Count of Participants; unit: Participants
Arm/Group | TSC 0.25 mg/kg - 9 Dose Group | TSC 0.25 mg/kg - 18 Dose Group
Number analyzed (Participants) | 3 | 0
Participants | 0 |

2. Primary Outcome: Overall Survival
Description: Participants in phase 2 (18 dose group, 6 weeks treatment with TSC) were monitored for up to 3 years (last follow-up - February 16, 2016). Overall Survival (OS) was defined as the length of time from the date of tumor resection surgery or definitive biopsy to the date of death. The OS analyses were performed using the Kaplan-Meier estimate method. The OS rates at 6, 12, 18 and 24 months were estimated. Median OS values were calculated; a corresponding 95% confidence interval for each median value was determined using a log rank analysis. The length of OS (in months) was calculated as follows: date of death or censored - date of surgery or definitive biopsy / 30.4375.
Time Frame: 6, 12, 18, 24 months
Population: All participants who received any amount of TSC and at least 1 session of RT (modified ITT)
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- TSC 0.25 mg/kg - 18 Dose Group - Phase 2: Trans Sodium Crocetinate (TSC): TSC administered intravenously for 18 doses as a bolus injection prior to radiation therapy sessions during 6 weeks of radiotherapy.
Arm/Group | TSC 0.25 mg/kg - 18 Dose Group - Phase 2
Number analyzed (Participants) | 56
participants
  6 month OS | 89.3 [81.18 to 97.39]
  12 month OS | 71.2 [59.22 to 83.09]
  18 month OS | 43.8 [30.67 to 56.90]
  24 month OS | 36.3 [23.55 to 49.08]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS analyses were performed using the Kaplan-Meier estimate method. The PFS rates at 6, 12, 18 and 24 months were estimated. Median PFS values were calculated; a corresponding 95% confidence interval for each median value was determined using a log rank analysis. Time to disease progression (in months) was calculated as follows: date of event* or censoring - date of surgery or definitive biopsy / 30.4375; *event = first tumor progression or death.
Time Frame: 6,12,18, 24 months
Population: The analysis of PFS was performed in phase 2 only and included the modified ITT population which included 54 of the 56 subjects (98.2%) at the 2-year time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TSC 0.25 mg/kg - 18 Dose Group - Phase 2
Number analyzed (Participants) | 56
percentage of participants
  6 months | 30.9 [18.70 to 43.12]
  12 months | 9.9 [1.80 to 18.03]
  18 months | 4.0 [0.00 to 9.32]
  24 months | 0.0 [0.00 to 0.00]

4. Secondary Outcome: Number of Participants With Reduction in Tumor Size, According to Percentage of Tumor Reduction
Description: The sum of the product of the diameters of the tumor (using recorded tumor diameter measurements made from brain MRI images) was used to express tumor size. Results were summarized for actual and percentage change from baseline. Individual subjects results were listed, including tumor volume and tumor response from independent reviewers. Investigator data were listed but not used in the analysis. Percent response (according to independent reviewer assessments) by percentage tumor reduction from tumor resection or definitive biopsy to the last MRI were summarized.
Time Frame: From Baseline to Week 110
Population: Of the 56 modified ITT population (subjects in the TSC 18 dose group) tumor size data exist for 37 subjects. Four (4) tumor-bearing subjects at baseline MRI did not have any post-baseline MRIs. Fourteen (14) subjects had a complete resection before baseline.
Measure: Count of Participants; unit: Participants
Groups:
- TSC 0.25mg/kg - 9 Dose Group - Phase 1: Phase 1 was the safety lead-in portion of the study conducted to evaluate an initial TSC dosage regimen in a smaller number of subjects and for a shorter period before a larger number of subjects were studied for a longer period in phase 2. Three (3) subjects were dosed with TSC at 0.25mg/kg for 3 weeks for a total of 9 doses with monitoring for dose-limiting toxicity (DLT). A Safety Monitoring Committee (SMC) evaluated the safety data and recommended TSC 0.25mg/kg for phase 2.
Arm/Group | TSC 0.25mg/kg - 9 Dose Group - Phase 1 | TSC 0.25 mg/kg - 18 Dose Group - Phase 2
Number analyzed (Participants) | 3 | 37
Participants
  tumor not reduced | 1 | 10
  0 to 39% tumor reduction | 0 | 6
  40 to 63% tumor reduction | 0 | 2
  64 to 93% tumor reduction | 0 | 6
  94 to 99% tumor reduction | 0 | 2
  100% tumor reduction | 2 | 11

ADVERSE EVENTS:
Time Frame: The first subject was enrolled February 27, 2012 and the last subject completed treatment on April 28, 2015. The last follow-up of the last subject was February 16, 2016. Adverse events were collected from the first dose of TSC to 30 days following the last dose (week 10 study visit). Subjects who experienced multiple events with the same preferred term were counted once for that preferred term.
Description: This was an open-label, sequential cohort, dose escalation study designed to evaluate the safety and efficacy of TSC administered concomitantly with standard-of-care RT and temozolomide in adults with GBM. The study included two phases. Phase 1 was a safety run-in wherein 3 subjects received 9 doses at 3 doses per week for 3 weeks. Phase 2 engaged 56 patients who received 18 doses at 3 doses per week for 6 weeks. The dose of TSC was consistently 0.25mg/kg.
Arm/Group | TSC 0.25 mg/kg - 9 Dose Group | TSC 0.25 mg/kg - 18 Dose Group
Serious Adverse Events (participants affected / at risk) | 1/3 | 10/56
Other Adverse Events (participants affected / at risk) | 3/3 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSC 0.25 mg/kg - 9 Dose Group (N=3) | TSC 0.25 mg/kg - 18 Dose Group (N=56)
Neutropenia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Brain edema (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSC 0.25 mg/kg - 9 Dose Group (N=3) | TSC 0.25 mg/kg - 18 Dose Group (N=56)
Fatigue (General disorders) | 0 (0) | 24 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 18 (20)
Nausea (Gastrointestinal disorders) | 0 (0) | 16 (17)
Constipation (Gastrointestinal disorders) | 0 (0) | 16 (16)
Headache (Nervous system disorders) | 0 (0) | 12 (13)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (13)
Insomnia (Psychiatric disorders) | 0 (0) | 9 (9)
Edema peripheral (General disorders) | 1 (1) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 7 (7)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (11)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (5)
Oral candidiasis (Infections and infestations) | 0 (0) | 5 (5)
Gait disturbance (General disorders) | 1 (1) | 3 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Confusional state (Psychiatric disorders) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Injection site bruising (General disorders) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (4)
Face edema (General disorders) | 0 (0) | 3 (3)
Irritability (General disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 3 (3)
Convulsion (Nervous system disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No